CLINICAL TRIAL: NCT06656624
Title: Efficacy and Safety of Ribociclib Combined With AI Versus Physician&Amp;#39;s Choice of Chemotherapy Sequential Endocrine Therapy in ER Medium to Low Expression/HER2-negative Advanced Breast Cancer: a Phase II Randomised Controlled Clinical Study
Brief Title: Efficacy and Safety of Ribociclib Combined With AI Versus Physician&Amp;#39;s Choice of Chemotherapy Sequential Endocrine Therapy in ER Middle-low-expression/HER2-negative Advanced Breast Cancer (Rachel)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Yidu Central Hospital of Weifang (Unknown); Affiliated Hospital of Jiangnan University (Other); The Affiliated Jiangyin Hospital of Southeast University Medical College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rachel
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Advanced Breast Cancer
Keywords: Ribociclib; ER medium to low expression; HER2 positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physician's choice of chemotherapy sequential Ribociclib combined with AI±OFS (Active Comparator)
  Interventions: Drug: physician's choice of chemotherapy sequential Ribociclib combined with AI±OFS
- Ribociclib combined with AI±OFS (Experimental)
  Interventions: Drug: Ribociclib combined with AI±OFS

INTERVENTIONS:
Drug: Ribociclib combined with AI±OFS — Ribociclib: 600mg /d, 3 weeks continuous oral withdrawal for 1 week; AI: Anastrozole 1mg, 1 time /d, oral; Letrozole: 2.5mg, 1 time /d, oral; Exemestane Tablets: 25mg, 1 time /d, oral Goserelin: 3.6 mg every 28 days, subcutaneous injection in the abdomen.
  Arms: Ribociclib combined with AI±OFS
Drug: physician's choice of chemotherapy sequential Ribociclib combined with AI±OFS — Docetaxel: 100mg/m2 IV drip every 21 days; Paclitaxel: 175mg/m2 every 21 days, IV drip; Paclitaxel for Injection (Albumin Bound): 100~150mg/m2 IV drip every 7 days; Capecitabine: 1000mg/m2, 2 times/d, 2 consecutive weeks of oral discontinuation for 1 week; Ribociclib: 600mg /d, 3 weeks continuous oral withdrawal for 1 week; AI: Anastrozole 1mg, 1 time /d, oral; Letrozole: 2.5mg, 1 time /d, oral; Exemestane Tablets: 25mg, 1 time /d, oral Goserelin: 3.6 mg every 28 days, subcutaneous injection in the abdomen.
  Arms: physician's choice of chemotherapy sequential Ribociclib combined with AI±OFS

SUMMARY:
To compare the efficacy and safety of ribociclib in combination with aromatase inhibitor and physician's choice of chemotherapy sequential endocrine therapy in the first-line treatment of ER medium to low expression/HER2-negative advanced breast cancer.

DETAILED DESCRIPTION:
The main goal of this clinical trial is to compare in the efficacy of Ribociclib in combination with AI versus physician's choice of chemotherapy sequential endocrine therapy in ER medium to low expression/HER2-negative advanced breast cancer and evaluate the PCR DFS,OS and safety of the subjects. The main question it aims is comparing the efficacy and safety of first-line application of CDK4/6 inhibitors combined with initial endocrine therapy versus sequential endocrine therapy after chemotherapy induction therapy in ER medium to low expression/HER2- negative advanced breast cancer.

This study is planned to include 190 patients with ER medium to low expression/HER2- negative advanced breast cancer between August 2024 and December 2025 who meet the entry criteria In this study, it is proposed to randomise the enrolled patients using stratified grouping + block randomisation method. The enrolled patients were firstly stratified based on (1) presence of visceral metastases and (2) disease-free interval ≤or ≥ 2 years assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is an adult female ≥ 18 years old at the time of informed consent.
2. ECGO rating 0-2.
3. Histologically confirmed recurrent or metastatic breast cancer, including patients initially diagnosed as stage IV or locally advanced inoperable patients.
4. Patient has a histologically and/or cytologically confirmed diagnosis of estrogen-receptor positive and/or progesterone receptor positive breast cancer based on the most recently analyzed tissue sample and all tested by local laboratory. ER should express in the range of 10% to 50%. ER positive by local laboratory testing.
5. Patient has HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1 + or 2 + If IHC is 2 +, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing and based on the most recently analyzed tissue sample.
6. Determination by the physician that the patient is in a rapid disease progression situation:

   * Symptomatic visceral metastases
   * Rapid progression of disease or impending visceral compromise.
   * Markedly symptomatic non visceral disease if the treating physician opt to give chemotherapy for rapid palliation of patients symptoms.
7. Patient hasn't received systemic anti-cancer therapy at the stage of recurrence/metastasis.
8. Patient must have at least one measurable lesion (according to RECIST 1.1 criteria)
9. Postmenopausal or pre/perimenopausal female patients are eligible for enrolment; pre or perimenopausal female patients must be willing to receive LHRHa during the study period.
10. All patients were required to meet the following laboratory biochemical values prior to enrolment:

    * Haematology: Hb ≥90 g/L, WBC ≥3.5×109/L, ANC ≥1.5×109/L, PLT ≥100×109/L;
    * Renal function: serum creatinine ≤ upper limit of normal value;
    * Liver function: for those without liver metastases, AST, ALT, ALP ≤2.5 times the upper limit of normal values, and ≤1.25 x the upper limit of normal values for total bilirubin; for those with liver metastases, AST, ALT, ALP ≤ 5 times the upper limit of normal value, and total bilirubin ≤ 1.5 x upper limit of normal value.

Exclusion Criteria:

1. Patient has received systemic anti-cancer therapy at the stage of recurrence/metastasis.
2. Those who have been treated with CDK4/6 inhibitors in the neoadjuvant/adjuvant phase.
3. Patients those with symptomatic CNS metastases.
4. Patient has a history of clinically symptomatic cardiovascular, hepatic, respiratory, renal and haemato-endocrine system or neuropsychiatric disorders.
5. Patient has a serious concomitant disease, such as an infectious disease; has multiple factors that affect the oral administration and absorption of the drug.
6. Pregnant or lactating women (women of childbearing age must have had a negative pregnancy test within 14 days prior to the first dose; if positive, pregnancy must be ruled out by ultrasound).
7. Patients in poor general condition who cannot tolerate chemotherapy treatment.
8. The investigator considers the patient unsuitable for entry into this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient is an adult female ≥ 18 years old at the time of informed consent.
Enrollment: 190 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression-free survival is defined as the time from the date of randomization to the date of the first documented progression as per local review and according to RECIST 1.1 or death due to any cause.the date of the first documented progression as per local review and according to RECIST 1.1 or death due to any cause.

SECONDARY OUTCOMES:
Progression Free Survival2 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Refers to the time from randomization to disease progression or death after a patient enters a clinical trial and receives second-line therapy.
Time to treatment failure | From randomization to treatment failure or withdrawal from the trial; reasons for withdrawal can be patient request, disease progression, death, or adverse events, whichever came first, assessed up to 100 months
  Time to treatment failure is defined as the time from the date of randomization/start of treatment to the earliest of date of progression, date of death due to any cause, change to other anti-cancer therapy, or date of discontinuation due to reasons other than 'Protocol violation' or 'Administrative problems'.
Overall response rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Overall response rate (ORR) is defined as the proportion of patients whose best overall response is either complete response (CR) or partial response (PR), as per local review and according to RECIST 1.1.
Overall survival(OS) | From date of randomization until the date of death from any cause, assessed up to 100 months
  Overall survival is defined as the time from the date of randomization to the date of death due to any cause.
Time To Response | From the date of randomization to the first documented response of either CR or PR, whichever came first, assessed up to 100 months
  Time to response is defined as the time from the date of randomization to the first documented response of either CR or PR, which must be subsequently confirmed, as defined by RECIST 1.1.
Clinical benefit rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Clinical benefit rate is defined as the proportion of patients with a best overall response of CR, or PR or stable disease, lasting for a duration of at least 24 weeks, as defined by RECIST 1.1.
Frequency/severity of adverse events | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Safety of ribociclib in combination with AI and OFS, and combination chemotherapies

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code